CLINICAL TRIAL: NCT03784937
Title: R-WITT Study : Revaluation of Wells' Clinical Prediction Score in Inpatients With Thromboprophylaxis Treatment
Brief Title: Revaluation of Wells' Clinical Prediction Score of Deep Vein Thrombosis (DVT) in Inpatients With Thromboprophylaxis Treatment
Acronym: R-WITT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 1994797v0; 2017-A02316-47 (Other: ANSM)
Record Dates: First submitted 2018-12-07; First posted 2018-12-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2018-12

CONDITIONS: Deep Vein Thrombosis; Thromboses, Venous
Keywords: Wells Clinical score; Thromboprophylaxis
MeSH Terms: conditions — Venous Thrombosis | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — Each patient received Doppler ultrasound for research of DVT, no matter the risk stratification.

SUMMARY:
This study aimed (1) revaluating the efficacy of the Wells' clinical prediction score for an inpatient population; and the weight of the presence of thromboprophylaxis treatment on the score, and (2) evaluating the correlation of a risk stratification established between a physician specialised in thrombosis and any other doctor.

ELIGIBILITY:
Inclusion Criteria:

* Any patient addressed to an Vascular Medicine unit for a clinical suspicion of DVT, with risk stratification through the modified Wells score by the referent doctor.

Exclusion Criteria:

* Patient addressed to our Vascular Medicine unit for any other reason.
* Patient addressed to our Vascular Medicine unit for DVT detection to help in a pulmonary embolism suspicion.
* Age under 18 yo
* Patients unable to express their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient adressed to an Vascular Medicine unit for a clinical suspicion of DVT, with risk stratification throught the modified Wells score by the referent doctor.
Sampling Method: Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Performance of the Wells Clinical prediction score | For enrollment to end of enrollment at 12 months
  Analyse area under the curve (AUC) of the Wells' score ROC (Receiver Operating Characteristic) curve for an inpatient population

SECONDARY OUTCOMES:
Impact of thromboprophylaxis treatment | For enrollment to end of enrollment at 12 months
  Compare area under curve of ROC curves of Wells' score between an inpatient population with or without thromboprophylaxis treatment
Coherency of Wells' score between an doctor specialized in thrombosis and any other doctor. | For enrollment to end of enrollment at 12 months
  Compare Area under curve for ROC curves of Wells' score between an doctor specialized in thrombosis and any other doctor.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalo-Universitaire de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trihan JE, Adam M, Jidal S, Aichoun I, Coudray S, Laurent J, Chaussavoine L, Chausserie S, Guillaumat J, Laneelle D, Perez-Martin A. Performance of the Wells score in predicting deep vein thrombosis in medical and surgical hospitalized patients with or without thromboprophylaxis: The R-WITT study. Vasc Med. 2021 Jun;26(3):288-296. doi: 10.1177/1358863X21994672. Epub 2021 Mar 22. PMID 33749393